CLINICAL TRIAL: NCT04229914
Title: Validity Reliability of 3 Meter Backward Walk Test in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ayşe Abit Kocaman, Principal investigator, Kırıkkale University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 3 Meter Backward Walk Test
Record Dates: First submitted 2020-01-01; First posted 2020-01-18 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Stroke Syndrome; Balance; Distorted; Walking, Difficulty
MeSH Terms: conditions — Stroke; Mobility Limitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stroke patients (Other): Assessment
  Interventions: Other: stroke patinets

INTERVENTIONS:
Other: stroke patinets — 3-m backwards walk test, timed up and go test, 10 m walk test, Berg BalanceTest, Functional Reach Test

SUMMARY:
The 3 m walk-back test is used to assess neuromuscular control, proprioception, protective reflexes, fall risk, and balance. In a study of healthy elderly adults, a 3-m walk-back test showed better diagnostic accuracy compared to the most commonly used measurement methods for falls in the past year. Reliability is extremely important, especially for research and clinical applications. In order to assess the risk of falling, measurement methods need to be reliable and change accurately over time. 3 m walk back test was found to be reliable in healthy elderly individuals. However, there are no studies investigating the validity and reliability of this test in stroke patients.

DETAILED DESCRIPTION:
Balance; within the limits of the stability of the center of gravity can be controlled on the surface. Balance can be affected due to muscle weakness after stroke, abnormal muscle tone, loss of deep sensation and disturbances in vestibular mechanisms. Among all sensorimotor results of stroke, it is stated that the balance of postural control has the greatest effect on daily living activities and gait. Accurate assessment of balance in stroke patients is important in identifying appropriate aids for mobility, choosing an effective treatment program, determining safe and unsafe activities, and setting rehabilitation goals. The most common risk factor for falls is one of the most important risk factors for stroke. Therefore, reliable and accurate measurement of dynamic gait balance is an important issue in stroke patients.The 3 m walk-back test is used to assess neuromuscular control, proprioception, protective reflexes, fall risk, and balance. In a study of healthy elderly adults, a 3-m walk-back test showed better diagnostic accuracy compared to the most commonly used measurement methods for falls in the past year. Reliability is extremely important, especially for research and clinical applications. In order to assess the risk of falling, measurement methods need to be reliable and change accurately over time. 3 m walk back test was found to be reliable in healthy elderly individuals. However, there are no studies investigating the validity and reliability of this test in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older,
* Getting a diagnosis of stroke,
* Not having cooperation and communication problems
* To be able to walk 10 m independently with or without device

Exclusion Criteria:

1. Have a neurological or orthopedic problem other than stroke that will affect functionality and balance
2. Individuals with contraindications for advanced cardiovascular disease and mobilization will not be included in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
3-m backwards walk test, | first day and second day
  A distance of 3 m is measured and marked with black tape. Individuals are asked to follow the heel and black band. With the 'start' command they are asked to walk backwards quickly. When the distance of 3 m is completed, a stop is instructed. Individuals are not allowed to run during the test. They are allowed to look back if they wish. The assessor walks behind individuals throughout the test. The test is repeated 3 times, the averages are recorded
timed up and go test | first day
  A standard chair is used for testing. First, the patient is asked to sit on the chair. The patient is then asked to stand up and walk regularly at a distance of 3 meters with a predetermined length, then return to the chair after 3 meters.
10 m walking test | first day
  In this test, the individual is asked to walk at his / her normal speed within a pre-measured 10-meter area and is started when the individual is at the starting line of the foot and terminated when he crosses the finish line.
Berg balance test | first day
  The BBS consists of 14 items to directly monitor the maintenance of body balance during performance.
Functional reach test | first day
  It is used to measure both the balance of the individual functionally and the amount of dynamic reach.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe A Abit Kocaman, Principal Investigator — Kırıkkale University
Locations (1):
- Ayşe Abit Kocaman, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carter V, Jain T, James J, Cornwall M, Aldrich A, de Heer HD. The 3-m Backwards Walk and Retrospective Falls: Diagnostic Accuracy of a Novel Clinical Measure. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):249-255. doi: 10.1519/JPT.0000000000000149. PMID 29095771